CLINICAL TRIAL: NCT02335697
Title: A Community-based Participatory Intervention to Change Attitudes Towards Female Circumcision Among Somali Immigrants in Sweden: a Cluster Randomized Controlled Trial
Brief Title: A Community-based Participatory Intervention to Change Attitudes Towards Female Circumcision Among Somali Immigrants in Sweden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Malmö University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Forte 2013-2095
Record Dates: First submitted 2015-01-07; First posted 2015-01-12 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Female Circumcision; Female Genital Mutilation/Cutting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Other): Attitude change towards female circumcision
  Interventions: Behavioral: Attitude change towards female circumcision
- No intervention (Other): No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Attitude change towards female circumcision — The intervention comprises of a series of meetings between newly arrived Somalis and established Somalis. At each meeting, a pre-determined topic relating to FC will be discussed. The topics include culture, religion, health, children's rights, and Swedish laws. Different experts, chosen to match the specific topic of the meeting will be invited to each meeting to facilitate the interactive discussions between the participants. Somalis who are both familiar with the Swedish and Somali culture will facilitate the meetings. The intervention spans over a time period of six months. The intervention meetings will be held during the first five months of the intervention period; one meeting scheduled per month. Thereafter, there will be a 'wash-out' period of one month to allow for reflections and to minimize the risk of courtesy bias.
  Arms: Intervention
Other: No intervention
  Arms: No intervention

SUMMARY:
Female circumcision (FC) causes both immediate and long-term health consequences. In general, the more severe type of FC, the worse health consequences can be seen. Despite the negative health effects, the practice of FC is still found to be highly prevalent in many countries, mainly in Africa and the Middle East. Many studies have been performed on FC in African countries where the custom is widespread and there have also been many attempts to eradicate the practice in these countries. However, considerably less research exists on FC in non-practicing societies where there has been an influx of immigrants from countries that traditionally carry out this practice. Further, no anti-FC interventions designed using a comparison group have been performed in any country outside Africa.

This cluster randomized controlled trial aims to evaluate the effectiveness of a community-based participatory intervention on changing attitudes towards FC among newly arrived Somali immigrants in Sweden. Included in the research is an assessment of the acceptability of the intervention. Based on social convention theory, we hypothesize that an interaction between established Somali immigrants, thought to be predominantly opponents of FC, and newly arrived Somali immigrants will facilitate changes in attitudes among the newly arrived.

The trial will be implemented in two municipalities in Sweden that have a high proportion of Somali immigrants. Somali organizations in these municipalities will constitute the clusters. In total, 8 clusters will be included, 4 intervention clusters and 4 control clusters.

ELIGIBILITY:
Inclusion Criteria:

* Oral informed consent
* Newly arrived (lived in Sweden for ≤ 4 years) Somali immigrants in Sweden with a residence permit
* Men and women, ≥ 18 years old

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) of types of female circumcision (change in what type of female circumcision the participant thinks is acceptable to do) | The outcome measure will be assessed before the intervention and approximately 1-30 days after the intervention.
  In the VAS, 0 mm indicates that no type of female circumcision is regarded as acceptable to do, and 100 mm indicates that all types of female circumcision are regarded as acceptable to do. The outcome will be the change in what type of female circumcision the participant thinks is acceptable to do, as measured by the change from the pre-intervention score.
Visual Analogue Scale (VAS) of types of female circumcision (change in what type of female circumcision the participant would perform if he/she had a daughter, as measured by the change from the pre-intervention score) | The outcome measure will be assessed before the intervention and approximately 1-30 days after the intervention.
  In the VAS, 0 mm indicates that the participant would not perform any type of female circumcision on his/her hypothesized daughter, and 100 mm indicates that the participant would perform the most extensive type of female circumcision on his/her hypothesized daughter. The outcome will be the change in what type of female circumcision the participant would perform if he/she had a daughter, as measured by the change from the pre-intervention score.
The change in proportion of participants who oppose the continuation of female circumcision | The outcome measure will be assessed before the intervention and approximately 1-30 days after the intervention

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) of types of female circumcision (participant assesses that Somali men in Sweden think that performing any type of female circumcision is not acceptable or acceptable) | The outcome measure will be assessed before the intervention and approximately 1-30 days after the intervention.
  In the VAS, 0 mm indicates that the participant assesses that Somali men in Sweden think that performing any type of female circumcision is not acceptable, and 100 mm indicates that the participant assesses that Somali men in Sweden think performing any type of female circumcision is acceptable. The outcome will be the change in the participant's assessment, as measured by the change from the pre-intervention score.
Visual Analogue Scale (VAS) of types of female circumcision (participant assesses that Somali women in Sweden think performing any type of female circumcision is acceptable or not acceptable) | The outcome measure will be assessed before the intervention and approximately 1-30 days after the intervention.
  In the VAS, 0 mm indicates that the participant assesses that Somali women in Sweden think performing any type of female circumcision is acceptable, and 100 mm indicates that the participant assesses that Somali women in Sweden think that performing all types of female circumcision is acceptable. The outcome will be the change in the participant's assessment, as measured by the change from the pre-intervention score.
Visual Analogue Scale (VAS) of number of individuals performing female circumcision | The outcome measure will be assessed before the intervention and approximately 1-30 days after the intervention.
  In the VAS, 0 mm indicates that the participant assesses that no one within the Somali community in Sweden circumcise their daughters, and 100 mm indicates that the participant assesses that everybody within the Somali community in Sweden circumcise their daughters. The outcome will be the change in the participant's assessment, as measured by the change from the pre-intervention score.
Change in answers to questions specifically related to one of the five topics of the intervention meetings | The outcome measures will be assessed before the intervention and approximately 1-30 days after the intervention.
Outcomes will be analyzed for associations with number of attended intervention meetings. | The outcome measure will be assessed approximately 1-30 days after the intervention.
Acceptability (questionnaire will be used to collect information about acceptability of the intervention) | The outcome measure will be assessed approximately 1-30 days after the intervention.
  A questionnaire will be used to collect information about acceptability of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta Essén, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

REFERENCES:
- [Derived] Wahlberg A, Johnsdotter S, Selling KE, Kallestal C, Essen B. Baseline data from a planned RCT on attitudes to female genital cutting after migration: when are interventions justified? BMJ Open. 2017 Aug 11;7(8):e017506. doi: 10.1136/bmjopen-2017-017506. PMID 28801440